CLINICAL TRIAL: NCT01041456
Title: Another Revisional Strategy to Address Severe Late Complications After Previous Biliopancreatic Diversion for Obesity: Major Revision From Standard Biliopancreatic Diversion to Proximal Roux-en-Y Gastric Bypass
Brief Title: Laparoscopic Revision From Biliopancreatic Diversion to Gastric Bypass
Acronym: BPD-to-RYGB
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Kelvin D Higa, MD, FACS; FASMBS; Professor of Surgery, University of California San Francisco, UCSF Fresno / ALSA Medical Group, Inc. Minimally Invasive Surgery Program
Other Study IDs: CMC IRB No. 2009016; U1111-1113-0264 (Other: World Health Organization, Universal Trial Number)
Record Dates: First submitted 2009-12-26; First posted 2009-12-31 (Estimated); Last update posted 2010-01-01 (Estimated); Status verified 2009-12

CONDITIONS: Metabolic and Nutritional Complications; Protein Malnutrition; Intestinal Malabsorptive Syndrome; Metabolic Bone Disease
Keywords: complicated biliopancreatic diversion; failed biliopancreatic diversion; revision gastric bypass; conversion bariatric surgery; revision bariatric surgery; re-operative bariatric surgery; malabsorptive syndrome; protein malnutrition; metabolic bone disease
MeSH Terms: conditions — Kwashiorkor; Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- complicated and/or failed BPD

SUMMARY:
The aim of this study is to describe the clinical presentation, indications, and operative treatment as well as assess the morbidity, mortality, and overall performance of revisional GBP after either failed and/or complicated Biliopancreatic Diversion "BPD" for weight loss. With such information, we hope to determine what features might assist us in advancing our knowledge about mechanisms of failure after primary bariatric surgery, mechanism of action of revisional GBP, and performance of revisional GBP through traditional outcome measurements as well as identifying predictors of good or poor outcome after revisional GBP in this specific subpopulation.

DETAILED DESCRIPTION:
In Italy, Professor Nicola Scopinaro, after studies in dogs, performed the first BPD in humans in 1976. Because of the lack of blind-loop syndrome and selective malabsorption for starch and fat, the BPD has an accepted risk-benefit ratio compared to the long ago abandoned Jejunoileal Bypass (a purely malabsorptive procedure). BPD side effects after resumption of full food intake include 2 to 4 bowel movements "BM" per day of foul-smelling, soft stools with flatulence. Modification of food habits and/or administration of neomycin or metronidazole for bacterial overgrowth syndrome tend to decrease BPD side effects after the disappearance of the postcibal syndrome somewhere around the fourth postoperative month.

To optimize its performance but mainly to decrease the protein malnutrition incidence, the BPD has undergone several modifications until 1992 when the ad hoc stomach-ad hoc alimentary limb BPD configuration was implemented. Consequently, the early sporadic and late recurrent forms of protein malnutrition have decreased from as high as 30% and 10% to as low as 2.0% and 1.0%, respectively.

PROTEIN-CALORIE MALNUTRITION

I) After BPD Protein-calorie malnutrition "PCM" is multifactorial and depends on patient-related factors (such as eating habits, capacity to adapt these to requirements set by the surgery, and socio-economic status) and technical factors (including gastric volume, bowel limb lengths, intestinal absorption and adaptation, and amount of endogenous nitrogen loss). Most cases are limited to a single or sporadic episode. In the early postoperative period secondary to the forced reduced food intake, the marasmic form of PCM incidence is higher, which is the aim of the operation. However, when carbohydrate intake is preferred (poor compliance with adequate protein intake), the hypoalbuminemic form will develop. The absorptive capacity of the alimentary limb "AL" and common limb or channel "CC" depends on 1) number of villi per square centimeter, 2) transit time, and 3) total intestinal length of the AL + CC. Thus, any condition that interferes with postoperative intestinal adaptation, mainly villous hypertrophy; increased transit time; and/or decreases the length of the functional AL + CC will lead to late onset of severe PCM. Increased number of bowel movements "BM" or severe diarrhea generally precedes to PCM.

After adequate counseling with life-style changes (mainly consumption of more than 90 g/day of high biological value protein), supplementation with pancreatic enzymes, and management of contributing medical conditions (such as gastroenteritis, lactose intolerance, intestinal bacterial overgrowth syndrome, celiac sprue, and inflammatory bowel disease), recurrent or severe PCM is frequently caused by excessive malabsorption. When mild or moderate protein malnutrition is instated, two to three weeks of parenteral nutrition are generally required to revert it. In contrast, severe PCM refers to the need for prolonged total parenteral nutrition "TPN", recurrent need for TPN, or malnutrition recalcitrant to TPN. Eventually, revisional surgery is required. The recurrent or severe form of PM is rarely secondary to excessive persistence of the food limitation mechanism with or without poor protein intake, requiring restitution of the intestinal continuity or complete reconstruction of the gastrointestinal tract (partial vs. full restoration). The partial restoration of the gastrointestinal tract allows normal protein-energy absorption, still partially preserving the specific effects of BPD on glucose and cholesterol metabolism.

II) After RYGB

1. Over a seven-year period, Avinoah et al. reported the nutritional status of 200 RYGB patients. Meat intolerance was observed in 51%, 60.3%, 59.5% and 55.1% of the patients during the 1st year, 2nd year, 3rd to 6th years, and 7th year after RYGB, respectively. No protein-calorie malnutrition was identified.
2. Moize et al. evaluated food consumption after 93 RYGB patients finding that inadequate protein intake is related to protein intolerance up to one year. Protein intake increased significantly over the first postoperative year from 45 g at 3 months, 46 g at 6 months, and to 58 g at 12 months. Low protein intake along the first year after RYGB is mainly related to intolerance to rich-protein food such as animal protein, mainly red meat.
3. There are no studies that quantify protein malabsorption after short-limb RYGB or any kind of RYGB variant. However, the less acidic environment of the gastric pouch after RYGB delays protein digestion by affecting the release of a cascade of peptides and enzymes, including pepsinogen, gastrin, and cholecystokinin which are involved in the initial breakdown of proteins.
4. In 236 consecutive short-limb, (6.3cm) banded RYGB patients, Faintuch et al. identified 4.7% patients with severe hypoalbuminemic malnutrition from which 63.6% had defined events, such as stenosis at the gastrojejunostomy (36.4%) or associated diseases, and 36.4% had severe emesis without any endoscopic abnormality.
5. In a series of 342 consecutive ringed RYGB, White et al. reported a 2% ring removal rate after placing a 6.5cm ring in 92 patients because of major restriction to solid foods.
6. In 65 patients converted to distal RYGB, Fobi et al. reported a mean BMI decrease of 7 kg/m2; however, 23% of patients developed protein malnutrition requiring revision surgery almost 50% of them.
7. In 27 distal RYGB at the 3rd postoperative year, Sugerman et al. reported a 25% incidence of protein malnutrition for the 150-cm common channel RYGB (n=22). In contrast, all five patients with a 50-cm common channel needed elongation of the common channel and two died of hepatic failure.

After extensive review of the literature, Kushner listed principal variables that contributed to nutritional deterioration after bariatric surgery: 1) sever malabsorption after malabsorptive procedures such as BPD or BPD-DS and distal or very, very long-limb RYGB; 2) surgical mechanical complications, such as stenosis at the gastrojejunostomy, intractable marginal ulcer, and gastro-gastric fistula; and 3) Non-compliance

Same analysis and review of the literature is available but less extensive for Metabolic bone disease, Anemia (Iron, folate, and vitamin B12), liposoluble vitamins and essential fatty acids.

Revisional strategies:

Revisional strategies that have been described for long-term complications after BPD are 1) elongation of common limb or channel, 2) restoration of intestinal continuity (partial restoration), and 3) restoration of gastrointestinal continuity (full restoration).

RYGB vs. BPD: Roux-en-Y configuration

1. Weight maintenance after BPD or BPD-DS appears to be superior to that after restrictive procedures and RYGB. However, this has never been subjected to a randomized controlled trial.
2. Intuitively, one would expect macro and micronutrient deficiency after bariatric surgery to be more frequent and severe when primarily malabsorptive with some restriction or pure malabsorptive procedures have been carried out, and this has been shown to be correct (level of evidence 3 or C).
3. Comparing the incidence rate of the largest series performed by experts, the incidence rate of late metabolic/nutritional complications after standard BPD/BPD-DS is higher than after standard RYGB.
4. There are trials with a level of evidence 3 & 4 (C & D) that favor the overall superiority of RYGB over BPD for clinically severe obesity including among others the following:

   * RYGB has been around longer than BPD
   * Widespread use of RYGB compared to BPD
   * Comparable weight loss however BPD has better weight maintenance than RYGB
   * RYGB has lower morbidity and mortality than BPD including metabolic/nutritional problems, which are more prevalent in BPD than in RYGB.
   * RYGB, in general, is accepted as the best revisional strategy for failed/ complicated restrictive procedures and even malabsortive surgeries such as the jejunoileal bypass

Summarizing, there is no evidence level A or 1 about what is the best overall primary bariatric procedure to address obesity at the long-term. In the USA, most investigators prefer RYGB for primary bariatric procedure, leaving BPD or BPD-DS for select cases including revisionary surgery for poor weight loss. After RYGB and BPD/BPD-DS, patients require to give priority for protein intake over other macronutrients as well as vitamin and mineral supplementation lifelong; there is no objective and standardized recommendation for supplementation. However, when metabolic/nutritional complications after BPD or BPD-DS develops regardless of optimized multispecialty medical management, lengthening of the common channel and partial or full reversals have been described. On the other hand, one-stage revision, either open or laparoscopic, from BPD to standard RYGB has never been reported. With this study, we will advance our knowledge about revisional RYGB, metabolic complications after hybrid bariatric procedures, and along with the existing literature, we will draw preliminary clinical recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Patients status post biliopancreatic diversion with any combination of the following severe late complications:

  * Metabolic and/or nutritional BPD-related complications.
  * Excessive weight loss
  * Poor weight loss, either Inadequate initial weight loss or Weight recidivism
  * Intolerable intestinal malabsorptive symptoms without severe malnutrition
* Undergoing either open or laparoscopic conversion to Roux-en-Y gastric bypass (RYGB) surgery.

Exclusion Criteria:

* Any other type of revision or conversion surgery.
* Adequate response to medical management of metabolic and nutritional complications after previous BPD
* missing records and/or unreachable patients with scant information for analysis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred with severe, persistent and/or recurrent metabolic/nutritional complications after open biliopancreatic diversion for clinically severe obesity underwent either laparoscopic or open conversion to Roux-en-Y gastric bypass. Intractability after interdisciplinary optimized medical therapy for metabolic and/or nutritional complications warranted surgical management.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2009-03; Primary Completion 2009-08 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Morbidity and mortality | at discharge, 1 week, 3 weeks, 8 weeks, 3 months, 6 months, 1 year and annually thereafter for up to 8 years
Weight loss expressed as Body Mass Index and Percentage of excess weight loss | at 6 months, 1 year and annually thereafter for up to 8 years

SECONDARY OUTCOMES:
Trend in comorbidities | at 6 months, 1 year, and annually thereafter for up to 8 years
Symptom resolution | at 6 months, 1 year, and annually thereafter for up to 8 years
Length of operative time which is defined as the time duration of operation measured in minutes from the first skin incision to the final closure of the skin incision | It is measured in minutes from the first skin incision to the final closure of the skin incision at the time of revisional surgery under study. It is a transoperative measure of outcome of the surgery under study
Length of Hospital Stay which is a measured of surgical recovery quantified and reported in days. It is a hospital pre-discharge traditional measure of outcome | It is measured in days from the admission date to the discharge date for the hospitalization pertaining to revisional surgery under study

CONTACTS AND LOCATIONS:
Overall Officials: Francisco M Tercero, MD, Study Director — Research Associate, University of California San Francisco; Kelvin D Higa, MD, Principal Investigator — Professor of Surgery, University of California San Francisco
Locations (1):
- UCSF Fresno Center for Medical Education and Research, Fresno, California, United States

REFERENCES:
- [Background] Higa KD, Boone KB, Ho T, Davies OG. Laparoscopic Roux-en-Y gastric bypass for morbid obesity: technique and preliminary results of our first 400 patients. Arch Surg. 2000 Sep;135(9):1029-33; discussion 1033-4. doi: 10.1001/archsurg.135.9.1029. PMID 10982506
- [Background] Hedley AA, Ogden CL, Johnson CL, Carroll MD, Curtin LR, Flegal KM. Prevalence of overweight and obesity among US children, adolescents, and adults, 1999-2002. JAMA. 2004 Jun 16;291(23):2847-50. doi: 10.1001/jama.291.23.2847. PMID 15199035
- [Background] McTigue KM, Harris R, Hemphill B, Lux L, Sutton S, Bunton AJ, Lohr KN. Screening and interventions for obesity in adults: summary of the evidence for the U.S. Preventive Services Task Force. Ann Intern Med. 2003 Dec 2;139(11):933-49. doi: 10.7326/0003-4819-139-11-200312020-00013. PMID 14644897
- [Background] Buchwald H, Avidor Y, Braunwald E, Jensen MD, Pories W, Fahrbach K, Schoelles K. Bariatric surgery: a systematic review and meta-analysis. JAMA. 2004 Oct 13;292(14):1724-37. doi: 10.1001/jama.292.14.1724. PMID 15479938
- [Background] Christou NV, Sampalis JS, Liberman M, Look D, Auger S, McLean AP, MacLean LD. Surgery decreases long-term mortality, morbidity, and health care use in morbidly obese patients. Ann Surg. 2004 Sep;240(3):416-23; discussion 423-4. doi: 10.1097/01.sla.0000137343.63376.19. PMID 15319713
- [Background] Adams TD, Gress RE, Smith SC, Halverson RC, Simper SC, Rosamond WD, Lamonte MJ, Stroup AM, Hunt SC. Long-term mortality after gastric bypass surgery. N Engl J Med. 2007 Aug 23;357(8):753-61. doi: 10.1056/NEJMoa066603. PMID 17715409
- [Background] Sjostrom L, Narbro K, Sjostrom CD, Karason K, Larsson B, Wedel H, Lystig T, Sullivan M, Bouchard C, Carlsson B, Bengtsson C, Dahlgren S, Gummesson A, Jacobson P, Karlsson J, Lindroos AK, Lonroth H, Naslund I, Olbers T, Stenlof K, Torgerson J, Agren G, Carlsson LM; Swedish Obese Subjects Study. Effects of bariatric surgery on mortality in Swedish obese subjects. N Engl J Med. 2007 Aug 23;357(8):741-52. doi: 10.1056/NEJMoa066254. PMID 17715408
- [Background] Cremieux PY, Buchwald H, Shikora SA, Ghosh A, Yang HE, Buessing M. A study on the economic impact of bariatric surgery. Am J Manag Care. 2008 Sep;14(9):589-96. PMID 18778174
- [Background] Santry HP, Gillen DL, Lauderdale DS. Trends in bariatric surgical procedures. JAMA. 2005 Oct 19;294(15):1909-17. doi: 10.1001/jama.294.15.1909. PMID 16234497
- [Background] Flum DR, Khan TV, Dellinger EP. Toward the rational and equitable use of bariatric surgery. JAMA. 2007 Sep 26;298(12):1442-4. doi: 10.1001/jama.298.12.1442. No abstract available. PMID 17895461
- [Background] Meguid MM, Glade MJ, Middleton FA. Weight regain after Roux-en-Y: a significant 20% complication related to PYY. Nutrition. 2008 Sep;24(9):832-42. doi: 10.1016/j.nut.2008.06.027. PMID 18725080
- [Background] Nguyen NT. Reoperations and revisions in bariatric surgery. Surg Endosc. 2007 Nov;21(11):1907-8. doi: 10.1007/s00464-007-9572-6. Epub 2007 Sep 8. No abstract available. PMID 17828427
- [Background] http://www.asbs.org/htm/Private/resolution.html. American Society of Metabolic and Bariatric Surgeons.
- [Background] Davies DJ, Baxter JM, Baxter JN. Nutritional deficiencies after bariatric surgery. Obes Surg. 2007 Sep;17(9):1150-8. doi: 10.1007/s11695-007-9208-x. PMID 18074487
- [Background] Brolin RE, Leung M. Survey of vitamin and mineral supplementation after gastric bypass and biliopancreatic diversion for morbid obesity. Obes Surg. 1999 Apr;9(2):150-4. doi: 10.1381/096089299765553395. PMID 10340768
- [Background] Scopinaro N, Gianetta E, Civalleri D, Bonalumi U, Bachi V. Bilio-pancreatic bypass for obesity: 1. An experimental study in dogs. Br J Surg. 1979 Sep;66(9):613-7. doi: 10.1002/bjs.1800660905. PMID 497644
- [Background] Scopinaro N, Gianetta E, Civalleri D, Bonalumi U, Bachi V. Bilio-pancreatic bypass for obesity: II. Initial experience in man. Br J Surg. 1979 Sep;66(9):618-20. doi: 10.1002/bjs.1800660906. PMID 497645
- [Background] Scopinaro N, Papadia F, Marinari G, et al. (2007). Biliopancreatic diversion. In Surgical Management of Obesity (pp.239-51). Philadelphia: Saunders.
- [Background] Scopinaro N, Marinari G, Camerini G, Papadia F; 2004 ABS Consensus Conference. Biliopancreatic diversion for obesity: state of the art. Surg Obes Relat Dis. 2005 May-Jun;1(3):317-28. doi: 10.1016/j.soard.2005.03.216. No abstract available. PMID 16925242
- [Background] Scopinaro N, Marinari GM, Pretolesi F, Papadia F, Murelli F, Marini P, Adami GF. Energy and nitrogen absorption after biliopancreatic diversion. Obes Surg. 2000 Oct;10(5):436-41. doi: 10.1381/096089200321594309. PMID 11054248
- [Background] Gianetta E, Friedman D, Adami GF, Vitale B, Traverso E, Castagnola M, Semino G, Scopinaro N. Etiological factors of protein malnutrition after biliopancreatic diversion. Gastroenterol Clin North Am. 1987 Sep;16(3):503-4. PMID 3125106
- [Background] Ren CJ. (2004). Laparoscopic malabsorption procedures: Complications. In Laparoscopic Bariatric Surgery (pp. 343-53). Philadelphia: Lippincott Williams & Wilkins.
- [Background] Scopinaro N, Gianetta E, Friedman D, Adami GF, Traverso E, Vitale B, Castagnola M, Semino G, Summa M, Bachi V. Surgical revision of biliopancreatic diversion. Gastroenterol Clin North Am. 1987 Sep;16(3):529-31. PMID 3436660
- [Background] Scopinaro N. Biliopancreatic diversion: mechanisms of action and long-term results. Obes Surg. 2006 Jun;16(6):683-9. doi: 10.1381/096089206777346637. No abstract available. PMID 16756725
- [Background] Scopinaro N. (2008). Biliopancreatic diversion: Revisional surgery. In obesity Surgery Principles and Practice (pp.277-83). New York: McGraw Hill.
- [Background] Avinoah E, Ovnat A, Charuzi I. Nutritional status seven years after Roux-en-Y gastric bypass surgery. Surgery. 1992 Feb;111(2):137-42. PMID 1736382
- [Background] Moize V, Geliebter A, Gluck ME, Yahav E, Lorence M, Colarusso T, Drake V, Flancbaum L. Obese patients have inadequate protein intake related to protein intolerance up to 1 year following Roux-en-Y gastric bypass. Obes Surg. 2003 Feb;13(1):23-8. doi: 10.1381/096089203321136548. PMID 12630609
- [Background] Ponsky TA, Brody F, Pucci E. Alterations in gastrointestinal physiology after Roux-en-Y gastric bypass. J Am Coll Surg. 2005 Jul;201(1):125-31. doi: 10.1016/j.jamcollsurg.2005.03.021. No abstract available. PMID 15978453
- [Background] Faintuch J, Matsuda M, Cruz ME, Silva MM, Teivelis MP, Garrido AB Jr, Gama-Rodrigues JJ. Severe protein-calorie malnutrition after bariatric procedures. Obes Surg. 2004 Feb;14(2):175-81. doi: 10.1381/096089204322857528. PMID 15018745
- [Background] White S, Brooks E, Jurikova L, Stubbs RS. Long-term outcomes after gastric bypass. Obes Surg. 2005 Feb;15(2):155-63. doi: 10.1381/0960892053268282. PMID 15802056
- [Background] Fobi MA, Lee H, Igwe D Jr, Felahy B, James E, Stanczyk M, Tambi J, Eyong P. Revision of failed gastric bypass to distal Roux-en-Y gastric bypass: a review of 65 cases. Obes Surg. 2001 Apr;11(2):190-5. doi: 10.1381/096089201321577866. PMID 11355025
- [Background] Sugerman HJ, Kellum JM, DeMaria EJ. Conversion of proximal to distal gastric bypass for failed gastric bypass for superobesity. J Gastrointest Surg. 1997 Nov-Dec;1(6):517-24; discussion 524-6. doi: 10.1016/s1091-255x(97)80067-4. PMID 9834387
- [Background] Kushner R. Managing the obese patient after bariatric surgery: a case report of severe malnutrition and review of the literature. JPEN J Parenter Enteral Nutr. 2000 Mar-Apr;24(2):126-32. doi: 10.1177/0148607100024002126. PMID 10772194
- [Background] Mazess RB, Barden HS, Drinka PJ, Bauwens SF, Orwoll ES, Bell NH. Influence of age and body weight on spine and femur bone mineral density in U.S. white men. J Bone Miner Res. 1990 Jun;5(6):645-52. doi: 10.1002/jbmr.5650050614. PMID 2382588
- [Background] Liel Y, Ulmer E, Shary J, Hollis BW, Bell NH. Low circulating vitamin D in obesity. Calcif Tissue Int. 1988 Oct;43(4):199-201. doi: 10.1007/BF02555135. PMID 3145124
- [Background] Coates PS, Fernstrom JD, Fernstrom MH, Schauer PR, Greenspan SL. Gastric bypass surgery for morbid obesity leads to an increase in bone turnover and a decrease in bone mass. J Clin Endocrinol Metab. 2004 Mar;89(3):1061-5. doi: 10.1210/jc.2003-031756. PMID 15001587
- [Background] Parfitt AM, Podenphant J, Villanueva AR, Frame B. Metabolic bone disease with and without osteomalacia after intestinal bypass surgery: a bone histomorphometric study. Bone. 1985;6(4):211-20. doi: 10.1016/8756-3282(85)90003-1. PMID 3840379
- [Background] Van Loan MD, Johnson HL, Barbieri TF. Effect of weight loss on bone mineral content and bone mineral density in obese women. Am J Clin Nutr. 1998 Apr;67(4):734-8. doi: 10.1093/ajcn/67.4.734. PMID 9537621
- [Background] Buffington C, Walker B, Cowan GS Jr, Scruggs D. Vitamin D Deficiency in the Morbidly Obese. Obes Surg. 1993 Nov;3(4):421-424. doi: 10.1381/096089293765559142. PMID 10757956
- [Background] Flancbaum L, Belsley S, Drake V, Colarusso T, Tayler E. Preoperative nutritional status of patients undergoing Roux-en-Y gastric bypass for morbid obesity. J Gastrointest Surg. 2006 Jul-Aug;10(7):1033-7. doi: 10.1016/j.gassur.2006.03.004. PMID 16843874
- [Background] Hamoui N, Anthone G, Crookes PF. Calcium metabolism in the morbidly obese. Obes Surg. 2004 Jan;14(1):9-12. doi: 10.1381/096089204772787211. PMID 14980026
- [Background] Ybarra J, Sanchez-Hernandez J, Gich I, De Leiva A, Rius X, Rodriguez-Espinosa J, Perez A. Unchanged hypovitaminosis D and secondary hyperparathyroidism in morbid obesity after bariatric surgery. Obes Surg. 2005 Mar;15(3):330-5. doi: 10.1381/0960892053576758. PMID 15826464
- [Background] Chapin BL, LeMar HJ Jr, Knodel DH, Carter PL. Secondary hyperparathyroidism following biliopancreatic diversion. Arch Surg. 1996 Oct;131(10):1048-52; discussion 1053. doi: 10.1001/archsurg.1996.01430220042009. PMID 8857901
- [Background] Bell NH, Greene A, Epstein S, Oexmann MJ, Shaw S, Shary J. Evidence for alteration of the vitamin D-endocrine system in blacks. J Clin Invest. 1985 Aug;76(2):470-3. doi: 10.1172/JCI111995. PMID 3839801
- [Background] Compston JE, Vedi S, Ledger JE, Webb A, Gazet JC, Pilkington TR. Vitamin D status and bone histomorphometry in gross obesity. Am J Clin Nutr. 1981 Nov;34(11):2359-63. doi: 10.1093/ajcn/34.11.2359. PMID 7304477
- [Background] Hey H, Stokholm KH, Lund B, Lund B, Sorensen OH. Vitamin D deficiency in obese patients and changes in circulating vitamin D metabolites following jejunoileal bypass. Int J Obes. 1982;6(5):473-9. PMID 6983505
- [Background] Riedt CS, Brolin RE, Sherrell RM, Field MP, Shapses SA. True fractional calcium absorption is decreased after Roux-en-Y gastric bypass surgery. Obesity (Silver Spring). 2006 Nov;14(11):1940-8. doi: 10.1038/oby.2006.226. PMID 17135609
- [Background] Johnson JM, Maher JW, DeMaria EJ, Downs RW, Wolfe LG, Kellum JM. The long-term effects of gastric bypass on vitamin D metabolism. Ann Surg. 2006 May;243(5):701-4; discussion 704-5. doi: 10.1097/01.sla.0000216773.47825.c1. PMID 16633006
- [Background] Allied Health Sciences Section Ad Hoc Nutrition Committee; Aills L, Blankenship J, Buffington C, Furtado M, Parrott J. ASMBS Allied Health Nutritional Guidelines for the Surgical Weight Loss Patient. Surg Obes Relat Dis. 2008 Sep-Oct;4(5 Suppl):S73-108. doi: 10.1016/j.soard.2008.03.002. Epub 2008 May 19. No abstract available. PMID 18490202
- [Background] Brolin RE, Gorman RC, Milgrim LM, Kenler HA. Multivitamin prophylaxis in prevention of post-gastric bypass vitamin and mineral deficiencies. Int J Obes. 1991 Oct;15(10):661-7. PMID 1752727
- [Background] Goode LR, Brolin RE, Chowdhury HA, Shapses SA. Bone and gastric bypass surgery: effects of dietary calcium and vitamin D. Obes Res. 2004 Jan;12(1):40-7. doi: 10.1038/oby.2004.7. PMID 14742841
- [Background] Johnson JM, Maher JW, Samuel I, Heitshusen D, Doherty C, Downs RW. Effects of gastric bypass procedures on bone mineral density, calcium, parathyroid hormone, and vitamin D. J Gastrointest Surg. 2005 Nov;9(8):1106-10; discussion 1110-1. doi: 10.1016/j.gassur.2005.07.012. PMID 16269381
- [Background] Youssef Y, Richards WO, Sekhar N, Kaiser J, Spagnoli A, Abumrad N, Torquati A. Risk of secondary hyperparathyroidism after laparoscopic gastric bypass surgery in obese women. Surg Endosc. 2007 Aug;21(8):1393-6. doi: 10.1007/s00464-007-9228-6. Epub 2007 Feb 21. PMID 17318692
- [Background] Marceau P, Biron S, Lebel S, Marceau S, Hould FS, Simard S, Dumont M, Fitzpatrick LA. Does bone change after biliopancreatic diversion? J Gastrointest Surg. 2002 Sep-Oct;6(5):690-8. doi: 10.1016/s1091-255x(01)00086-5. PMID 12399058
- [Background] Hamoui N, Kim K, Anthone G, Crookes PF. The significance of elevated levels of parathyroid hormone in patients with morbid obesity before and after bariatric surgery. Arch Surg. 2003 Aug;138(8):891-7. doi: 10.1001/archsurg.138.8.891. PMID 12912749
- [Background] Newbury L, Dolan K, Hatzifotis M, Low N, Fielding G. Calcium and vitamin D depletion and elevated parathyroid hormone following biliopancreatic diversion. Obes Surg. 2003 Dec;13(6):893-5. doi: 10.1381/096089203322618722. PMID 14738677
- [Background] Slater GH, Ren CJ, Siegel N, Williams T, Barr D, Wolfe B, Dolan K, Fielding GA. Serum fat-soluble vitamin deficiency and abnormal calcium metabolism after malabsorptive bariatric surgery. J Gastrointest Surg. 2004 Jan;8(1):48-55; discussion 54-5. doi: 10.1016/j.gassur.2003.09.020. PMID 14746835
- [Background] Dolan K, Hatzifotis M, Newbury L, Fielding G. A comparison of laparoscopic adjustable gastric banding and biliopancreatic diversion in superobesity. Obes Surg. 2004 Feb;14(2):165-9. doi: 10.1381/096089204322857500. PMID 15018743
- [Background] DeMaria EJ. Is gastric bypass superior for the surgical treatment of obesity compared with malabsorptive procedures? J Gastrointest Surg. 2004 May-Jun;8(4):401-3. doi: 10.1016/j.gassur.2003.12.022. No abstract available. PMID 15120361
- [Background] Dolan K, Hatzifotis M, Newbury L, Lowe N, Fielding G. A clinical and nutritional comparison of biliopancreatic diversion with and without duodenal switch. Ann Surg. 2004 Jul;240(1):51-6. doi: 10.1097/01.sla.0000129280.68540.76. PMID 15213618
- [Background] Brolin RE, Gorman JH, Gorman RC, Petschenik AJ, Bradley LB, Kenler HA, Cody RP. Prophylactic iron supplementation after Roux-en-Y gastric bypass: a prospective, double-blind, randomized study. Arch Surg. 1998 Jul;133(7):740-4. doi: 10.1001/archsurg.133.7.740. PMID 9688002
- [Background] Brolin RE, LaMarca LB, Kenler HA, Cody RP. Malabsorptive gastric bypass in patients with superobesity. J Gastrointest Surg. 2002 Mar-Apr;6(2):195-203; discussion 204-5. doi: 10.1016/s1091-255x(01)00022-1. PMID 11992805
- [Background] Marceau P, Hould FS, Lebel S, Marceau S, Biron S. Malabsorptive obesity surgery. Surg Clin North Am. 2001 Oct;81(5):1113-27. doi: 10.1016/s0039-6109(05)70187-0. PMID 11589248
- [Background] Brolin RE, Gorman JH, Gorman RC, Petschenik AJ, Bradley LJ, Kenler HA, Cody RP. Are vitamin B12 and folate deficiency clinically important after roux-en-Y gastric bypass? J Gastrointest Surg. 1998 Sep-Oct;2(5):436-42. doi: 10.1016/s1091-255x(98)80034-6. PMID 9843603
- [Background] Halverson JD. Micronutrient deficiencies after gastric bypass for morbid obesity. Am Surg. 1986 Nov;52(11):594-8. PMID 3777703
- [Background] Marcuard SP, Sinar DR, Swanson MS, Silverman JF, Levine JS. Absence of luminal intrinsic factor after gastric bypass surgery for morbid obesity. Dig Dis Sci. 1989 Aug;34(8):1238-42. doi: 10.1007/BF01537272. PMID 2666054
- [Background] Skroubis G, Sakellaropoulos G, Pouggouras K, Mead N, Nikiforidis G, Kalfarentzos F. Comparison of nutritional deficiencies after Roux-en-Y gastric bypass and after biliopancreatic diversion with Roux-en-Y gastric bypass. Obes Surg. 2002 Aug;12(4):551-8. doi: 10.1381/096089202762252334. PMID 12194550
- [Background] Rhode BM, Tamin H, Gilfix BM, Sampalis JS, Nohr C, MacLean LD. Treatment of Vitamin B12 Deficiency after Gastric Surgery for Severe Obesity. Obes Surg. 1995 May;5(2):154-158. doi: 10.1381/096089295765557953. PMID 10733805
- [Background] Ocon Breton J, Perez Naranjo S, Gimeno Laborda S, Benito Ruesca P, Garcia Hernandez R. [Effectiveness and complications of bariatric surgery in the treatment of morbid obesity]. Nutr Hosp. 2005 Nov-Dec;20(6):409-14. Spanish. PMID 16335025
- [Background] Boylan LM, Sugerman HJ, Driskell JA. Vitamin E, vitamin B-6, vitamin B-12, and folate status of gastric bypass surgery patients. J Am Diet Assoc. 1988 May;88(5):579-85. PMID 3367015
- [Background] Mechanick JI, Kushner RF, Sugerman HJ, Gonzalez-Campoy JM, Collazo-Clavell ML, Guven S, Spitz AF, Apovian CM, Livingston EH, Brolin R, Sarwer DB, Anderson WA, Dixon J. American Association of Clinical Endocrinologists, The Obesity Society, and American Society for Metabolic & Bariatric Surgery Medical Guidelines for Clinical Practice for the perioperative nutritional, metabolic, and nonsurgical support of the bariatric surgery patient. Surg Obes Relat Dis. 2008 Sep-Oct;4(5 Suppl):S109-84. doi: 10.1016/j.soard.2008.08.009. Epub 2008 Aug 19. PMID 18848315
- See also: "Click here for more information about the department sponsor´s web site" — http://www.fresno.ucsf.edu/surgery/